CLINICAL TRIAL: NCT06965660
Title: Prevalence and Burden of Balance Disorders in Community-dwelling Older Adults: A Population-based Study Protocol
Brief Title: Population Cohort Set-up for the Epidemiological Assessment of Balance Disorders in Elderly People
Acronym: EPIBAS
Status: Active, not recruiting | Type: Observational
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Karolinska Institutet (Other); Fundació Tecnocampus Mataró-Maresme (Other); Fundació Institut Germans Trias i Pujol (Other); Universidade da Coruña (Other)
Responsible Party: Principal Investigator, Pilar Montero Alía, Bachelor of Medicine and Surgery. PhD medicine., Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Other Study IDs: PI20/00406; PI20/00406 (Other Grant/Funding Number: Instituto de Salud Carlos III)
Record Dates: First submitted 2025-04-10; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-04

CONDITIONS: Balance Disorders; Accidental Falls; Frailty; Aging
Keywords: Postural balance; Balance disorders; Falls; Posturography; Retinal microvasculature; Nintendo Wii Balance Board™; Knee extensor strength; Aging; Prevalence; Health Assessment Tool (HAT); Cognitive function; Epidemiology
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Age-based cohort of people aged 65-75 living in Mataró, Spain: Eligibility criteria:
  * Aged 65-75.
  * Reside in Mataró.
  * Able to walk independently, with or without technical assistance.
  Exclusion criteria:
  * Unable to walk independently.
  * Terminal illness or severe cognitive decline.
  * Incompetence in Catalan or Spanish.
  * Lack of phone access

SUMMARY:
As people age, it becomes more common to experience balance problems. These issues can increase the risk of falling, which may lead to serious health consequences and loss of independence. While many studies have looked at falls in older adults, there is still limited information about how many people actually have balance disorders, how these disorders develop over time, and which factors might help detect them early-before a fall happens.

This clinical study aims to understand how common balance disorders are among older adults aged 65 to 75, how they change over time, and which simple, accessible tools might help us predict who is at risk. The study will include over 1,300 participants living in Mataró (Barcelona, Spain), who will be followed for a period of 18 months.

Participants will undergo a series of assessments to measure their balance, leg strength, and general health. One key test is posturography, an advanced method that evaluates how well a person can maintain balance. In addition, the study will explore the use of a simple tool-the Nintendo Wii™ Balance Board-as a low-cost way to detect balance issues. Retinal photographs will also be taken to study the small blood vessels in the eye, which may reflect changes in brain circulation that affect balance. Lastly, a tool called the Health Assessment Tool (HAT) will be used to assess participants' overall physical and cognitive function.

The study hypothesizes that certain indicators-such as leg strength, changes in retinal blood vessels, balance performance using tools like the Wii™, and overall health assessments (HAT)-can help predict who is at greater risk for balance problems and falls. The study also explores whether posturography, as a gold-standard method, can reveal how balance disorders are related to the risk and consequences of falling.

Detecting balance problems early can help prevent falls, reduce the risk of injury, and support older adults in maintaining their independence. This study may help identify easy and effective methods to screen for balance disorders, improving quality of life for older adults and reducing the personal and healthcare costs associated with falls.

DETAILED DESCRIPTION:
Background:

Poor balance leads to falls, which can result in loss of personal autonomy and reduced quality of life. Epidemiological studies on balance disorders (BDs) remain scarce. It is essential to determine the prevalence and incidence of BDs and to identify potential markers that facilitate their detection and monitoring in an accessible and practical way.

Aims:

* To assess the prevalence of BDs in men and women aged 65-72 using posturography and a variety of balance tests, and to monitor the annual incidence of BDs.
* To analyze the relationship between retinal microvasculature abnormalities and balance impairments.
* To evaluate the effectiveness of the Wii Balance Board™ as a tool for balance assessment compared to posturography.
* To explore whether knee extensor strength and a composite measure of physical and cognitive function can serve as predictors of BDs and fall risk.
* To externally validate the Health Assessment Tool (HAT scale) in the Spanish population.

Methods:

This is a two-phase observational study.

* Phase I: Descriptive, cross-sectional.
* Phase II: Cohort follow-up at 18 months. A total of 1,316 individuals aged 65-75 residing in Mataró (Barcelona, Spain) will be included, excluding those unable to walk independently. Participants will undergo posturography, retinal imaging, knee extensor strength measurement, and a battery of functional tests: Tinetti Test, Timed Up and Go test, Unipedal Stance Test, Short Physical Performance Battery (SPPB), and balance assessment using the Nintendo Wii at baseline and at the end of follow-up. Bimonthly phone calls will be conducted to detect fall events.

Applicability and relevance:

BDs are often underdiagnosed and undertreated. Current awareness of the problem is limited. Enhancing knowledge in this field is crucial to prevent the loss of functional autonomy and to develop targeted preventive strategies for those at highest risk of falls. This will allow for a more efficient and evidence-based approach to this prevalent geriatric syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65-75.
* Reside in Mataró.
* Able to walk independently, with or without technical assistance.

Exclusion Criteria:

* Unable to walk independently.
* Terminal illness or severe cognitive decline.
* Incompetence in Catalan or Spanish.
* Lack of phone access.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The target population is an age-based cohort of people aged 65-75 living in Mataró. This age range was selected to find individuals who do not yet have BDs, enabling the calculation of the incidence. According to the 2017 municipal register, and the population's age structure, there are 2,215 people in this age range. A total of 1,316 people will be randomly selected to form a sample stratified by gender and age from the Primary Care Information System (SIAP) database, which includes health cardholders. The SIAP is not as exhaustive or up-to-date as the population census. This register includes any individual ascribed to a primary care center (covering nearly the entire population), regardless of whether or not they have used this health service and whether they are healthy or ill. Our research team will contact the selected participants using the phone number registered in the SIAP and invite them to take part in the study.
Sampling Method: Probability Sample
Enrollment: 1300 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Posturography | Baseline and 18-month follow-up
  Static posturography measures the displacement of the center of pressure while standing on a force platform. Greater sway indicates poorer balance control. Also looks at dynamic stability.
  The balance assessment is based on the comparison of the parameters that best discriminate the pathology of the general population with those obtained from patterns of normality segmented by age (database of the Institute of Biomechanics of Valencia). Ratings are displayed in percentages, so that results other than 100% reflect discrepancy with respect to normal values. It is considered pathological when the results are less than 95%, indicating that these subjects are more likely to present an alteration in the studied system. Pathological values for the limits of stability are considered to be below 85%.
Unipedal Stance Test | Baseline and 18-month follow-up
  The test measures whether the participant is able to stand on one leg without support for 5 seconds.
Timed Up and Go (TUG) Test | Baseline and 18-month follow-up
  Time in seconds taken to rise from a chair, walk 3 meters, turn around, return, and sit down again. Shorter times indicate better functional mobility and lower fall risk.
Tinetti Test | Baseline and 18-month follow-up
  The Tinetti assesses gait and balance. It consists of two components: balance (maximum 16 points) and gait (maximum 12 points), for a total score ranging from 0 to 28 points. Higher scores indicate better balance and gait performance, and lower risk of falls.
Short Physical Performance Battery (SPPB) | Baseline and 18-month follow-up
  The Short Physical Performance Battery is an objective tool for measuring functional capacity, balance, and lower limb strength in adults over 65 years old. The test includes three different domains to assess functional mobility: gait, sit-to-stand, and balance. A score below 8 indicates mobility and physical exercise limitations and is associated with a higher risk of mobility disability and, consequently, a higher risk of falls. A score of 8 or higher is considered within the normal range.
Balance Assessment Using the Nintendo Wii Console | Baseline and 18-month follow-up
  This includes the test of the gimp leg and center of gravity assessment, as well as Romberg Test variants: Eyes Open (REO), Eyes Closed (REC), and on Foam Pad (RuFP), as performed in the posturography test. The Nintendo Wii provides accurate measures of body center of pressure (COP), an important metric for balance stability assessment approximating the body's center of mass. The Romberg test assesses gait disturbance caused by abnormal proprioception, disequilibrium from central vertigo, and peripheral vertigo. Patients is asked to stand with feet together, arms next to the body, first with eyes open and then closed. The patient tries to maintain his balance. The test is scored by counting the seconds the patient can stand with eyes closed.
Muscle Strength of Lower Limbs | Baseline and 18-month follow-up
  Measurement of force in kilograms of the lower extremities using a hand-held dynamometer or similar device. Higher values indicate greater muscle strength
Gait Speed | Baseline, 6-month follow-up, and 18-month follow-up
  Measurement of usual walking speed (in seconds) over a distance of 6 meters. Higher speeds indicate better functional mobility.
Physical activity measured using the abbreviated Spanish version of the Minnesota Leisure-Time Physical Activity Questionnaire (VREM) | Baseline and 18-month follow-up
  The VREM is a short version in Spanish of the Minnesota Leisure Time Physical Activity Questionnaire (CAFM). It is a tool designed to assess the quality and quantity of physical activity performed during leisure time. It consists of 6 items that evaluate the physical activity performed in the last month, taking into account only the activities performed during free time.
  The energy expenditure is quantified in MET-min/14 days by multiplying the METs of each physical activity by its duration (in minutes) by the frequency accumulated in the month prior to the interview and by the months of the year in which the activity was performed. Furthermore, it is divided by 365 days/year and multiplied by 14 days. Then, it is classified according to the energetic cast:
  * Very active: Energy index higher than 5,000 METs-min/14 days.
  * Active: Energy index between 3,000 and 4,999 METs-min/14 days.
  * Moderately active: Energy index between 1,250 and 2,999 METs-min/14 days.
  * Sedentary: Energy index
Lawton-Brody Instrumental Activities of Daily Living (IADL) | Baseline, 6-month follow-up, and 18-month follow-up
  The scale evaluates complex daily activities (e.g., cooking, managing finances). Scores range from 0 (low function, dependent) to 8 (high function, independent). Higher scores indicate better functional capacity.
Barthel Index of Activities of Daily Living (ADL) | Baseline, 6-month follow-up, and 18-month follow-up
  Assesses performance in basic activities such as bathing, dressing, and feeding. Scores range from 0 to 100. Higher scores indicate greater independence.

SECONDARY OUTCOMES:
Health Assessment Tool (HAT) | 6-month follow-up
  Health status will be assessed using the Health Assessment Tool (HAT), a composite measure integrating the following five health dimensions:
  1. Physical function, assessed by gait speed (measured over 4 meters);
  2. Cognitive function, assessed by the Mini-Mental State Examination (MMSE), ranging from 0 to 30, with higher scores indicating better cognitive function;
  3. Chronic morbidity, determined by the number of diagnosed chronic conditions recorded using the ICD-10 classification system;
  4. Mild disability, assessed using the Lawton-Brody Instrumental Activities of Daily Living (IADL) scale, excluding household tasks to reduce gender bias;
  5. Severe disability, assessed using the Barthel Index for basic activities of daily living (ADLs), focusing on five essential self-care tasks (bathing, toileting, transferring, eating, and dressing).
  These dimensions will be combined to generate a composite health status profile, according to the HAT methodology.
Retinography | Baseline and 18-month follow-up
  Retinal images will be analyzed to assess microvascular parameters using two software tools:
  1. IMEDOS Vessel Map software (IMEDOS Systems UG, Germany) will be used to measure retinal vessel diameters and calculate central retinal arteriolar equivalent (CRAE), central retinal venular equivalent (CRVE), and arteriolar-to-venular ratio (AVR).
  2. SIRIUS software (University of A Coruña) will be used to calculate retinal vessel tortuosity and arteriovenous (A/V) ratio.
  These parameters serve as non-invasive biomarkers of microvascular health.

OTHER OUTCOMES:
Short Falls Efficacy Scale - International (Short FES-I) | Baseline and 18-month follow-up
  Fear of falling will be assessed using the Short Falls Efficacy Scale - International (Short FES-I), a 7-item self-reported questionnaire that evaluates concern about falling during basic daily activities. Each item is rated from 1 (not at all concerned) to 4 (very concerned), yielding a total score from 7 to 28. Higher scores indicate greater fear of falling.
History of Falls | Every 2 months from baseline through month 18 (i.e., at months 0, 2, 4, 6, 8, 10, 12, 14, and 18)
  Participants will self-report the number of falls experienced in the 12 months preceding study enrollment, along with fall-related consequences (e.g., injuries, fractures, hospitalizations). The variable includes both quantitative (number of falls) and qualitative (presence of consequences) components.
Charlson Comorbidity Index | Baseline and 18-month follow-up
  Comorbidity will be assessed using the Charlson Comorbidity Index (CCI), a validated method for classifying prognostic comorbidity in longitudinal studies. The CCI assigns weighted scores based on the presence of 17 predefined chronic conditions.
  Additionally, the total number of chronic conditions and specific ICD-10 diagnoses recorded in the patient's electronic health record will be documented.
Mini-Mental State Examination (MMSE) | Baseline and 18-month follow-up
  Cognitive function will be assessed using the MMSE, a 30-item scale. Total scores range from 0 to 30, with higher scores indicating better cognitive function.
Pfeiffer Short Portable Mental State Questionnaire (SPMSQ) | Baseline
  Cognitive impairment will be assessed using the SPMSQ, a 9-item scale. Scores range from 0 to 9 errors. Scores greater than 5 errors indicate moderate to severe cognitive impairment.
UCLA-3 Loneliness Scale | Baseline or 18-month follow-up
  Perceived loneliness will be assessed using the 3-item UCLA Loneliness Scale (UCLA-3), which evaluates subjective feelings of social isolation and lack of companionship. Each item is scored from 1 (hardly ever) to 3 (often), for a total score ranging from 3 to 9. Higher scores indicate greater loneliness.
De Jong Gierveld Loneliness Scale | Baseline or 18-month follow-up
  Loneliness will also be assessed using the De Jong Gierveld Loneliness Scale, a validated 6-item questionnaire that distinguishes between emotional and social loneliness. Items are scored and interpreted following the official scoring algorithm, with higher scores indicating greater loneliness.
Blood Sample | Baseline
  Blood samples will be collected from participants for future analysis of biomarkers related to frailty and sarcopenia. The collected samples will be stored for use in subsequent studies aimed at identifying and validating relevant biomarkers.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina - USR Metropolitan North., Mataró, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No